CLINICAL TRIAL: NCT04299945
Title: The Effects of Dietary Nitrate Supplementation on Exercise Tolerance in Patients With Fibrotic Interstitial Lung Disease
Brief Title: Effects of Drinking Beetroot Juice on Exercise Performance in Patients With Fibrotic Interstitial Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Director of Cardiopulmonary Exercise Physiology Laboratory, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H19-02552
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Interstitial Lung Disease
Keywords: ILD; Nitrates; exercise; interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial; Motor Activity

STUDY DESIGN:
Intervention Model Description: One or more interventions are evaluated for maximizing comfort, minimizing side effects, or mitigating against a decline in the participant's health or function
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomly assigned using a computer-generated algorithm in a 1:1 ratio to dietary nitrate supplementation (concentrated beetroot juice) or placebo (the same amount of beetroot juice but with naturally occurring nitrate removed).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary nitrate supplementation (Experimental): The dietary nitrate supplement will be a concentrated, nitrate-rich beetroot juice (70 ml providing ∼400mg nitrate per serving)
  Interventions: Dietary Supplement: concentrated beetroot juice (400mg of nitrate per serving)
- Placebo (Placebo Comparator): The placebo will be a concentrated, nitrate-depleted beetroot juice (70 ml with trace amounts of nitrate)
  Interventions: Dietary Supplement: concentrated beetroot juice (trace amounts of nitrate per serving)

INTERVENTIONS:
Dietary Supplement: concentrated beetroot juice (400mg of nitrate per serving) — Dietary nitrate supplementation includes consumption of two beverages daily for 7 consecutive days.
  Arms: Dietary nitrate supplementation
Dietary Supplement: concentrated beetroot juice (trace amounts of nitrate per serving) — Dietary placebo supplementation includes consumption of two beverages daily for 7 consecutive days.
  Arms: Placebo

SUMMARY:
Exercise training as part of a structured pulmonary rehabilitation program is a key factor in improving quality of life and symptoms in people with interstitial lung disease (ILD). Optimal methods of exercise training are yet to be explored in ILD. Drinking beetroot juice, which is rich in nitrate, has been shown to improve exercise performance in a variety of groups, but its effects in ILD have not been tested. The purpose of this study is to determine if drinking nitrate-rich beetroot juice can improve exercise performance compared to drinking nitrate-free beetroot juice in people with ILD.

DETAILED DESCRIPTION:
PURPOSE:

The primary purpose of this study is to determine the effects of dietary nitrate supplementation on submaximal cycle exercise performance in patients with fibrotic ILD.

HYPOTHESIS:

Our primary hypothesis is that dietary nitrate supplementation will result in greater improvement in submaximal cycle exercise endurance time compared with placebo.

JUSTIFICATION:

Fibrotic interstitial lung disease (ILD) is a heterogeneous group of disorders that cause scarring/fibrosis or inflammation of the lungs, resulting in significant morbidity and high mortality. Almost all ILDs are characterized by dyspnoea and functional limitation and there are few effective and/or well-tolerated pharmacotherapies for many ILD subtypes.

Exertional dyspnoea leads to reduced exercise capacity in ILD, and this functional limitation is further worsened by skeletal muscle weakness and dysfunction. Both dyspnoea and poor exercise tolerance are strongly associated with quality of life and mortality in ILD and thus improving dyspnoea and functional capacity are important goals in the management of ILD.

Pulmonary rehabilitation is a structured evidence-based exercise and education intervention that is recommended for most patients with ILD. Pulmonary rehabilitation improves dyspnoea, functional capacity, and quality of life in patients with ILD; however, these benefits are often modest and only temporary. The exercise component of pulmonary rehabilitation is the predominant mediator of benefit; however, there are no studies that have investigated the optimal method of exercise training in patients with ILD. Thus, there is a clear need to identify new strategies that can provide larger and more persistent benefits from pulmonary rehabilitation.

Nitric oxide (NO) is a physiological signaling molecule that plays a critical role in vascular control. There is accumulating evidence that dietary nitrate, consumed in the form of beetroot juice, can increase the bioavailability of NO and subsequently enhance exercise performance in healthy, elite athlete, as well as diseased populations. These improvements may be related, but not limited to, enhanced efficiency of locomotion, peripheral locomotor oxygen delivery, and/or muscle power. The specific effects of dietary nitrate supplementation in ILD patients has yet to be explored. However, there is great potential for the use of this dietary supplement to improve exercise tolerance during, and improve patient outcomes from, pulmonary rehabilitation.

STATISTICAL ANALYSIS:

A p value <0.05 will be considered significant for all analyses. Data analysis will be performed using Microsoft Excel 2013 (Microsoft Corporation, Redmond, Washington, US) and Stata v12 (StataCorp, Texas, US).

Primary outcome: The primary outcome of cycle endurance time will be based on the duration patients were able to exercise during the constant work rate exercise test. A t-test will be used to compare endurance times between the intervention and placebo conditions.

The investigators have chosen to power this study based on the primary outcome of change in cycle exercise endurance time. Based on previously collected data in our laboratory in patients with ILD that show a standard deviation of 289.96 seconds for a 75% constant work rate cycle exercise test with a conservative between test correlation of 0.90, the investigators calculated that 15 participants would be needed to detect the minimal clinically important difference of 105 seconds between conditions assuming a two-sided α of 0.05 and 80% power.

ELIGIBILITY:
Inclusion Criteria:

* A multidisciplinary diagnosis of idiopathic pulmonary fibrosis (IPF), idiopathic fibrotic nonspecific interstitial pneumonia (NSIP), chronic hypersensitivity pneumonitis (HP), or unclassifiable ILD with a differential diagnosis that consists of the above diagnoses
* Fibrosis on high resolution computed tomography (HRCT): honeycombing, reticulation, or traction bronchiectasis
* Oxygen saturation ≥92% by pulse oximetry at rest while breathing room air
* Clinically stable for the preceding 6 weeks
* Can fluently read and write in English

Exclusion Criteria:

* Contraindication to exercise testing (e.g. significant cardiovascular, musculoskeletal, neurological disease) (see Table 4 from ERS/ATS consensus statement)
* Other significant pulmonary or extra-pulmonary disease that, based on clinical assessment, could impair exercise capacity and/or oxygenation
* FVC <50% or DLCO <25%
* Use of prednisone >10 mg/day for >2 weeks within 3 months of the first study visit
* Cardiac pacemaker or any metal or electronics inside of the body

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in submaximal cycle exercise endurance time following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Exercise endurance time will be measured during submaximal constant load cycle exercise testing.

SECONDARY OUTCOMES:
Difference in exertional dyspnoea during submaximal cycle exercise following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Dyspnea rating, measured using the Borg 0-10 category ratio scale, will be assessed at rest and every 1 minute during submaximal constant load cycle exercise testing until exhaustion.
Difference in exertional dyspnoea during activities of daily living following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Shortness of breath during daily living patterns will be assessed using established questionnaires.
Difference in concentration of plasma nitrate ([NO3-]) and nitrite ([NO2-]) following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Blood samples will be taken and analyzed for the concentration levels of nitrates in blood plasma.
Difference in resting, exercise, and post-exercise blood pressure following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Blood pressure will be measured using a manual sphygmomanometer at rest, every 2 minutes during submaximal constant load cycle exercise testing until exhaustion, and 5 minutes after exercise ends.
Difference in oxygen cost of submaximal cycle exercise following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Oxygen consumption will be measured during submaximal constant load cycle exercise testing.
Difference in peripheral locomotor muscle oxygenation following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Peripheral locomotor muscle oxygenation will be monitored using near-infrared spectroscopy during submaximal constant load exercise testing.
Difference in post-exercise quadriceps fatigue following dietary nitrate supplementation compared to placebo supplementation. | 1 Week
  Quadriceps fatigue will be assessed by measuring the quadriceps muscle force output using the femoral magnetic stimulation technique immediately before and after submaximal constant load exercise testing.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Providence Health Care - St. Paul's Hosptial, Vancouver, British Columbia
  - Vancouver Coastal Health, Vancouver

IPD SHARING:
Plan to Share IPD: No